CLINICAL TRIAL: NCT03987100
Title: Population Pharmacokinetics of Amoxicillin in Neonates: Evaluation and Optimization of the Dose
Brief Title: Population Pharmacokinetics of Amoxicillin in Neonates
Acronym: NEOPOPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18-9874
Record Dates: First submitted 2019-01-09; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood or cerebrospinal fluid drawn for routine biochemical tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of NEOPOPI is to conduct a population pharmacokinetic study of amoxicillin in neonates, in order to evaluate and optimize neonatal dose regimen.

There will be no change to the medication treatment received by participants. An opportunistic pharmacokinetic sampling approach will be followed: samples will be scavenged from blood or cerebrospinal fluid drawn for routine biochemical tests. In this way, no additional invasive tests will be needed.

DETAILED DESCRIPTION:
* Administration of the antibiotic according to the usual procedures for prescribing services: in particular, neither the indications nor the doses nor the methods of administration are fixed by the protocol
* Opportunistic sampling strategy: no biological samples are specifically collected for the purposes of the study (measurements of concentrations on "bottoms" or "left-over" samples); the performance of this non-invasive sampling strategy has been previously demonstrated in the neonatal population.
* Micro-analytical method (assay of concentrations on micro-volumes, of the order of 50μL)
* Population pharmacokinetic analysis

ELIGIBILITY:
Inclusion Criteria:

* Neonates receiving amoxicillin and blood/CSF tests during amoxicillin treatment, as part of their routine clinical care
* No parental opposition to the study participation

Exclusion Criteria:

• None

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (including both preterm and full-term neonates) receiving amoxicillin as part of their routine clinical care (for suspected or proven neonatal sepsis).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of therapeutic efficacy target of amoxicillin | 1 week
  Achievement rate of therapeutic efficacy target of amoxicillin (ie percentage of neonates in whom amoxicillin plasma concentration remains above the MIC of target organisms for more than 70% of the dose range). In accordance with the recommendations of the European Medicines Agency, the optimal dosage regimen is defined as leading to a probability of antibiotic therapy success of greater than or equal to 90%. Thus, it is necessary to determine the dosage regimen allowing the target of therapeutic efficacy to be reached (ie maintenance of the plasma concentration of amoxicillin greater than the MIC of the targeted microorganisms for more than 70% of the dose) in at least 90% of treated neonates.

SECONDARY OUTCOMES:
Recording of Adverse Events | 1 week
  Recording of adverse events (clinical and / or biological) during the treatment period and up to 96 hours after the end of treatment
Minimum Inhibitory Concentration | 1 week
  Collection of MICs of amoxicillin for isolated germs. For amoxicillin the antibacterial activity is time-dependent, the predictor of efficacy is the "Time> MIC": this is the percentage of the administration interval during which the concentration of the antibiotic remains higher than the MIC of target germs
Concentration of amoxicilin in Cerebrospinal Fluid (CSF) | 1 week
  Calculation of amoxicillin concentration in CSF / amoxicillin plasma concentration when data permits (i.e. when lumbar puncture is performed as part of usual care, during treatment with amoxicillin

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France